CLINICAL TRIAL: NCT07251218
Title: A Cluster Randomised Controlled Trial (cRCT) Evaluating the Effects of Cool Roofs on Mental Health Outcomes in Ahmedabad, India
Brief Title: Assessing the Effects of Cool Roofs on Mental Health in Ahmedabad, India
Acronym: REFLECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aditi Bunker (Other)
Collaborators: Heidelberg University (Other); Rutgers University (Other); Boston University (Other); Indian Institute of Public Health, India (Other); Sika (Unknown); University of Auckland, New Zealand (Other)
Responsible Party: Sponsor-Investigator, Aditi Bunker, Co-principal investigator, University of Auckland, New Zealand
Organization: University of Auckland, New Zealand (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3728166; 226745/Z/22/Z (Other Grant/Funding Number: Wellcome Trust UK)
Record Dates: First submitted 2025-11-13; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Eco-anxiety; PTSD - Post Traumatic Stress Disorder; Resilience; Anxiety
Keywords: Cool roof; Mental health; Heat stress; Housing; Hot temperature; Humidity
MeSH Terms: conditions — Combat Disorders; Anxiety Disorders; Psychological Well-Being; Heat Stress Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Trial participants will be aware of the intervention to which they have been allocated, and the research fieldworkers will be aware of the intervention allocation. The trial steering committee members and trial statistician will remain blinded until the end of trial period and data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cool roof (Experimental): Households will receive sunlight reflecting 'cool roof' coating on their roofs.
  Interventions: Other: Cool roof
- No cool roof (No Intervention): No cool roof application. Households will keep their original roofing for the duration of the trial.

INTERVENTIONS:
Other: Cool roof — Cool roofs are a heat-reflecting material that can be applied to existing household roofing in the form of a liquid-applied membrane. Cool roofs work by increasing solar reflectance (the ability to reflect the visible wavelengths of sunlight, reducing heat transfer to the surface) and thermal emittance (the ability to radiate absorbed solar energy) thereby reducing the amount of heat transferred into the home.
  Arms: Cool roof

SUMMARY:
Ambient air temperatures in India have broken record highs. Solutions are needed to build heat resilience in communities and adapt to increasing heat from climate change. Sunlight-reflecting cool roof coatings may passively reduce indoor temperatures and energy use to protect home occupants from extreme heat. Occupants living in poor housing conditions are susceptible to increased heat exposure.

Heat exposure can instigate and worsen mental health. The worst adverse health effects are experienced in communities that are least able to adapt to heat exposure. By reducing indoor temperatures, cool roof use can promote mental wellbeing in household occupants.

The long-term research goal of the investigators is to identify viable passive housing adaptation technologies with proven health benefits to reduce the burden of heat stress in communities affected by heat. To meet this goal, the investigators will conduct a cluster-randomized controlled trial to establish the effects of cool roof use on mental health in Ahmedabad, India.

DETAILED DESCRIPTION:
Increasing heat exposure from climate change is causing and exacerbating heat-related illnesses in millions worldwide - particularly in low resource settings. June 2024 was the 13th consecutive hottest month on record globally - shattering previous records. Heat exposure can instigate and worsen mental health conditions, including depression, anxiety and aggression. Adaptation is essential for protecting people from increasing heat exposure. The built environment, especially homes, are ideal for deploying interventions to reduce heat exposure and accelerate adaptation efforts. However, there currently is a lack of evidence on a global scale - generated through empirical studies - guiding the uptake of interventions to reduce heat stress in low resource settings.

Sunlight-reflecting cool roof coatings passively reduce indoor temperatures and lower energy use, offering protection to home occupants from extreme heat. The investigators therefore aim to conduct a cluster-randomized controlled trial investigating the effects of cool-roof use on mental health outcomes in Ahmedabad.

The trial will quantify whether cool roofs are an effective passive home cooling intervention with beneficial health effects for vulnerable populations in Ahmedabad. Findings will inform regional policy responses on scaling cool roof implementation to protect people from increasing heat exposure driven by climate change.

ELIGIBILITY:
Inclusion Criteria:

* Permanent household resident.

Exclusion Criteria:

* Roof damage, inaccessible or instability of roof adversely affecting cool roof coating application.
* Participant unable to provide written/verbal informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Depression | Eight measurements will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Self-reported presence and frequency of symptoms of depression assessed using aggregate score of the Patient Health Questionnaire 9 (PHQ-9). Minimum score of 0 and a maximum score of 27 with a higher score meaning a worse outcome.

SECONDARY OUTCOMES:
Aggression | Eight measurements: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Self-reported personal aggresion assessed using the Buss-Perry Aggression Questionnaire-Ultra Short Form (BPAQ-ML).
Mental Well-being | One measurement at the end of follow-up at 12 months post-intervention
  Self-reported mental wellbeing over the last two weeks using the Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS) with a minimum score of 14 and a maximum score of 70. A higher score indicates a higher level of mental well-being.
Resilience | One measurement at the end of follow-up at 12 months post-intervention.
  Self-reported resilience rating over the last month using the Connor-Davidson Resilience Scale (CD-RISC-10) with a minimum score of 0 and a maximum score of 40. Higher total scores indicate a greater ability to cope with adversity and higher resilience.
Eco-anxiety | One measurement taken at the end of follow-up at 12 months post-intervention.
  Self-reported eco-anxiety over the last two weeks measured using the Hogg Eco-Anxiery Scale with a total score range from a minimum of 0 to a maximum of 52. Higher scores on the scale and its sub-dimensions indicate higher levels of eco-anxiety.
Post-Traumatic Stress Disorder | One measurement taken at the end of follow-up at 12 months post-intervention.
  Self-reported symptoms of post-traumatic stress disorder using the Short PTSD Rating Interview (SPRINT) questionnaire with a potential score range from a minimum of 0 to a maximum of 32. A higher score indicates greater PTSD symptoms.
Anxiety | One measurement at the end of follow-up at 12 months post-intervention.
  Self-reported anxiety over the last two weeks using the GAD-7 Anxiety Severity Scale with a minimum score of 0 and a maximum score of 21. Higher scores indicate greater anxiety severity.

CONTACTS AND LOCATIONS:
Overall Officials: Collin Tukuitonga, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- IndianI Institute of Public Health Gandhinagar, Ahmedabad, India

IPD SHARING:
Plan to Share IPD: Yes
Data that can be shared unconditionally underpinning the published research articles will be made available to other researchers at the time of publication, and data will be linked via the article DOI. Data that cannot be unconditionally shared upon publication owing to confidentiality or data protection requirements will be identified as such and a contact email will be provided in relevant publications for data access enquiries by other researchers. Individual names of study participants and identifying factors will be removed prior to data sharing.
  It is expected that demographic data of people at the study sites (family size and composition, basic socioeconomic indicators) may contain personally identifiable information and location data. All such data will be removed prior to storage on online data repositories and therefore will be available to be publicly shared at the time of publication of manuscripts.
Supporting Information: ICF, CSR
Time Frame: At the time of publication.
URL: http://reflect.org.nz